CLINICAL TRIAL: NCT06221007
Title: Evaluation of Long-Term Results of Bone Cement Application in Stapes Surgery and Factors Effective on Results in Stapes Surgery
Brief Title: Long-Term Results of Bone Cement in Stapes Surgery
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof Dr, Pamukkale University
Other Study IDs: 17
Record Dates: First submitted 2024-01-13; First posted 2024-01-24 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Otosclerosis
Keywords: stapedotomy; otosclerosis
MeSH Terms: conditions — Otosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Use of bone cement in otosclerosis surgery — Surgical technique; It involves separating the sclerosed stapes from the oval window and incus under an endoscope or microscope and replacing it with a Teflon piston, which is a middle ear prosthesis. In this way, a new connection between the incus and the oval window ensures the transmission of sound to the inner ear. Bone cement has long been used in primary and revision ossiculoplasty, including stapedotomy of the middle ear. During stapedotomy, the part of the Teflon piston that places the teflon piston on the incus is fixed with bone cement, aiming to keep the prosthesis in place for a long time and prophylactic treatment of incus necrosis.

SUMMARY:
Considering the long-term results of otosclerosis surgery performed in our clinic, it was observed that in addition to the improvement in air conduction hearing, which indicates conductive hearing, which is the main success of the surgery, there was also an improvement in bone conduction hearing, which indicates sensorineural hearing, in patients using bone cement.

Our study aimed to examine the effect of bone cement use in otosclerosis surgery on long-term hearing thresholds and bone conduction.

DETAILED DESCRIPTION:
A retrospective review was conducted on records of patients who underwent stapes surgery between 2012 and 2020.

Comprehensive records were selected, and patients were summoned for clinic visits for thorough examinations. Evaluation encompassed the average of air and bone conduction at 500, 1000, 2000, and 4000 Hz. A procedure-specific 16-item questionnaire and the Glasgow Benefit Inventory (GBI) were used for perceived benefit and effective factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 who underwent stapedotomy with a diagnosis of otosclerosis

Exclusion Criteria:

* Inadequate information in files

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Stapedotomy surgeries performed at Pamukkale University ENT clinic since 2011 will be examined retrospectively.
Sampling Method: Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Incidence of improvement of conductive hearing loss in patients using bone cement | through study completion, an average of 7 year
  Changes in conductive hearing loss will be examined using pure tone audiometry testing.

SECONDARY OUTCOMES:
Incidence of decrease in bone conduction hearing threshold in patients using bone cement | through study completion, an average of 7 year
  The change in sensorineural hearing threshold will be examined using pure tone audiometry test.
Glasgow Benefit inventory | through study completion, an average of 7 year
  The GBI is an 18-item, validated instrument designed specifically to assess patient-perceived benefits following otolaryngologic interventions. It utilizes a five-point Likert scale. The score is changing between -100(worst) and +100(best). Total scores interpreted as follows: >50 indicates significant benefit, 10-50 indicates moderate benefit, and <10 denotes no perceived benefit.
Postoperative questinarie | through study completion, an average of 7 year
  16 items stapedotomy specific questions

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No